CLINICAL TRIAL: NCT04343846
Title: Eruption Status of Primary Teeth and BMI in Low Birth Weight Children in Comparison to Normal Birth Weight Children
Brief Title: Eruption Status of Primary Teeth in Low Birth Weight Children in Comparison to Normal Birth Weight Childern
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Magdy Sayed Mohamed, principal investigator, Cairo University
Other Study IDs: primary teeth eruption
Record Dates: First submitted 2020-02-19; First posted 2020-04-13 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-01

CONDITIONS: Eruption Statues of Primary Teeth in LBW Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: low birth weight children
- group B: normal birth weight children

SUMMARY:
determine the status of eruption of primary teeth and physical growth in children aged from 6 to 36 months with low birth weight in comparison to normal birth weight

DETAILED DESCRIPTION:
Timing of eruption of primary teeth is an urgent question for every mother especially in low birth weight children. Although, the timing of eruption of primary teeth and their sequence of eruption shown to be under the genetic control , pre-natal maternal conditions, early childhood metabolic and nutritional factors along with socioeconomic states have been associated with the timing of eruption of primary teeth.

Many factors may affect the timing of eruption. Literature showed that factors like gender, race and physical growth may influence emergence of tooth in child mouth but there is scarce information on Egyptian children .

ELIGIBILITY:
Inclusion Criteria:

* Healthy children.
* Children aged from 6 to 36 month.

Exclusion Criteria:

* Refusal of participation from the parents.
* Medically compromised children.
* Major illness.
* The child had special needs.
* Any systemic disease.
* Any congenital deformity that may affect teeth eruption.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children aged from 6 months to 36 months
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
status of eruption of primary teeth | 1 year
  clinical examination

SECONDARY OUTCOMES:
child physical growth | 1 year
  weight in kilograms height in centimeter weight and height will be combined to report BMI in kg/m^2

REFERENCES:
- [Background] Shaweesh AI, Al-Batayneh OB. Association of weight and height with timing of deciduous tooth emergence. Arch Oral Biol. 2018 Mar;87:168-171. doi: 10.1016/j.archoralbio.2017.12.030. Epub 2017 Dec 29. PMID 29304424
- [Background] Soliman NL, El-Zainy MA, Hassan RM, Aly RM. Relationship of deciduous teeth emergence with physical growth. Indian J Dent Res. 2012 Mar-Apr;23(2):236-40. doi: 10.4103/0970-9290.100433. PMID 22945716